CLINICAL TRIAL: NCT00324259
Title: A Phase II Randomized Study of Physiological (6 mg Daily) and High Dose (30 mg Daily) Estradiol in the Treatment of Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Study of Physiological and High Dose Estradiol in the Treatment of Hormone Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0412 / 201108392
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (6 mg estradiol) (Active Comparator): 6 mg of estradiol daily (2 mg tid).
  Interventions: Drug: Estradiol
- Arm 2 (30 mg estradiol) (Active Comparator): 30 mg of estradiol. (10 mg tid)
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol

SUMMARY:
This study aims to examine whether estradiol is an appropriate for future Phase 3 studies as second or third line endocrine treatment. In addition the protocol explores several approaches to enhance the safety of estrogen therapy, including the establishment of the efficacy of a lower dose than that currently recommended and through the early identification of non-responders to avoid drug exposure in patients who are unlikely to benefit to estrogen treatment.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of two doses (6 mg and 30 mg) of Estradiol, a type of estrogen. This and other forms of estrogen used at doses much higher than those used for postmenopausal hormone replacement therapy have been shown to cause tumor growth stabilization or shrinkage in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with advanced hormone receptor positive (ER and or PgR) breast cancer, has received prior treatment with an aromatase inhibitor in the advanced disease setting, and experienced at least 24 weeks of progression free survival. As long as the patient experienced an aromatase inhibitor response as defined this way, she is still eligible even if she has received further lines of endocrine therapy, which may include other aromatase inhibitors or tamoxifen, even if these subsequent lines of treatment were unsuccessful (see below for permitted chemotherapy and trastuzumab therapy).

OR

* Postmenopausal women with systemic or unresectable local relapse after taking at least two years of adjuvant aromatase inhibitor therapy.
* Clinical diagnosis of postmenopausal status is defined as either:

  1. Age greater than 50 years and amenorrhea for 1 year
  2. Bilateral Surgical ovariectomy
  3. Serum FSH and estradiol level in the postmenopausal range before the initiation of AI therapy.
  4. If the patient was receiving an LHRH agonist to maintain a postmenopausal state during AI therapy this should be continued since recovery of menses would lead to uncontrolled estrogen exposure and pregnancy during estrogen therapy is contraindicated.
* Tumor cell expression of ER and/or PgR can be ascertained on either the primary or the metastatic site. However when both types of tissue are available, the metastatic site should be used to determine eligibility. ER and/or PgR positive are defined as at least 10% of malignant cells with positive nuclear staining.
* The patients may have received adjuvant and/or neoadjuvant chemotherapy.
* Prior radiotherapy is permitted as long as it was planned before the start of the study medication and is completed within 3 weeks of trial medication starting.
* Prior tamoxifen therapy is also permitted as adjuvant or advanced disease therapy.
* Patients with ER+ HER2+ disease are eligible even of they have received trastuzumab in the past (and even if it was administered in combination with endocrine treatment) as long as they meet all other eligibility criteria. Trastuzumab therapy must be held during estradiol treatment.
* Use of prior experimental agents alone or in combination with endocrine therapy is also permissible, but a wash out of one month is required if the immediate prior therapy involved a study medication that had not been subject to regulatory approval.
* Prior adjuvant chemotherapy is permitted as well as one line of chemotherapy for advanced disease.
* Patient must have at least one measurable lesion defined by RECIST criteria. To be considered measurable, a baseline lesion must have a minimum diameter to compensate for measurement error: 1 cm for soft tissue lesions, 1 cm for lung lesions including pleural lesions measured by CT scan, 1 cm for liver lesions measured by CT scan.
* Patients with bone only disease can also be enrolled if they meet the following criteria:

  1. Four or more lesions more than one cm, measurable on CT scan bone windows.
  2. At least one tumor marker that is elevated to at least two times the upper limit of normal.
  3. All patients should have a baseline bone scan with X-ray evaluation of all hot spots, CT chest abdomen and pelvis (with bone windows), and tumor marker assessment. Also CT scan of the extremities should be done on suspicious areas seen on X-ray evaluation of all hot spots if these extremity lesions are to be followed for response.
* The patient must have an ECOG performance status of 0-2
* The patient should have a life expectancy of > 6 months.
* The patient must have adequate hematologic function, defined as ANC >1000/mm3 and platelets > 75,000/mm3.
* The patient must have adequate renal function, defined as serum creatinine less than or equal to 1.5 times the upper limit of normal.
* The patient must have adequate liver function defined as serum bilirubin less than or equal to 1.5 times the upper limit of normal (three times the upper limit of normal for patients with hereditary benign hyperbilirubinaemia), transaminases (ALT, AST) less than or equal to 2.5 times the upper limit of normal in patients without liver metastasis or less than or equal to 5 times the upper limit of normal in patients with liver metastasis.
* For patients with bone metastasis, treatment with i.v. bisphosphonates during the trial is mandatory because of the risk of hypercalcemia. Bisphosphonate therapy must be started before the patient begins protocol therapy.
* Preexisting hypercalcemia should be treated and calcium normalized prior to study entry.
* The patient must give written informed consent prior to initiation of any invasive study-related procedures that would otherwise not be performed, and must be able to comply with scheduled visits and evaluations.
* Inclusion of Women and Minorities: Entry to this study is open to women of all racial and ethnic subgroups.
* Patients with fasting blood glucose level ≤ 200 mg/dL. If greater, hyperglycemia must be treated before initiation of study investigations.

Exclusion Criteria:

* Patients with CNS involvement with metastatic breast cancer or life threatening lymphangitic or large volume lung or liver disease that threatens organ function.
* Patients with history of deep venous thrombosis, pulmonary embolism, stroke, acute myocardial infarction, congestive cardiac failure, untreated hypertension.
* Ischemic changes on a baseline EKG or other evidence of ischemic heart disease.
* Undiagnosed abnormal genital bleeding
* Untreated cholelithiasis
* Fasting serum triglycerides greater than 400. Patients should be treated and triglycerides controlled prior to study entry.
* Treatment with fulvestrant within 12 months of study initiation (fulvestrant has been shown to antagonize estradiol induced apoptosis in preclinical models (5).
* The patient's only qualifying lesion (s) have been previously irradiated or are scheduled for irradiation following study entry.
* Severe or uncontrolled concomitant disease from other causes.
* EGOG Performance status 3 or 4.
* The patient has previous malignancies other than breast cancer except a) adequately treated in situ carcinoma of the cervix, b) localized basal or squamous cell carcinoma of the skin c) any previous malignancy treated with curative intent with a recurrence risk of less than 30%.
* The patient is unable to understand the informed consent or is unlikely to be compliant with the protocol.
* More than one line of palliative chemotherapy for advanced disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-08; Primary Completion 2011-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ellis, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina Breast Clinic, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western University, Cleveland, Ohio
  - Cleveland Clinic, Lerner College of Medicine, Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Ellis MJ, Gao F, Dehdashti F, Jeffe DB, Marcom PK, Carey LA, Dickler MN, Silverman P, Fleming GF, Kommareddy A, Jamalabadi-Majidi S, Crowder R, Siegel BA. Lower-dose vs high-dose oral estradiol therapy of hormone receptor-positive, aromatase inhibitor-resistant advanced breast cancer: a phase 2 randomized study. JAMA. 2009 Aug 19;302(7):774-80. doi: 10.1001/jama.2009.1204. PMID 19690310
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/03/2004 and closed to participant enrollment on 02/19/2008.
Period: Overall Study
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol) | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Median (Full Range); unit: years] | 54.7 [36.3 to 83.8] | 59.5 [39.4 to 77.7] | 57.1 [36.3 to 83.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 66
Site [Number; unit: participants]
  Bone/soft tissue | 18 | 13 | 31
  Visceral | 5 | 5 | 10
  Both | 11 | 14 | 25
Estrogen receptor status [Number; unit: participants]
  Negative | 1 | 0 | 1
  Positive | 33 | 32 | 65
Progesterone receptor status [Number; unit: participants]
  Negative | 8 | 6 | 14
  Positive | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CR Plus PR Plus SD)
Description: Complete response (CR) + partial response (PR) + stable disease (SD) using RECIST 1.0
  CR = disappearance of all target lesions
  PR = at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter
  SD = neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for progressive disease
  SD is defined as lack of disease progression by 24 weeks.
Time Frame: 24 weeks after start of treatment
Measure: Number; unit: participants
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 34 | 32
participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 3 | 1
  Stable disease (SD) | 7 | 8
  CR+PR+SD | 10 | 9

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from treatment initiation to disease progression or death.
  Time of last observation for patients remaining in the study and the time at which dose reductions, study drug termination, and withdrawal of consent occurred were treated as censored data.
  Indicated as number of participants who had not progressed at 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Progression per RECIST 1.0 = at least a 20% increase in the sum of the longest diameter of target lesions taking as references the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 48 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 34 | 32
participants
  12 weeks (no progression) | 30 | 20
  24 weeks (no progression) | 13 | 9
  36 weeks (no progression) | 7 | 6
  48 weeks (no progression) | 6 | 3

3. Secondary Outcome: Quality of Life
Description: Surveyed using a 6 item estrogen adverse effect questionnaire (headaches, bloating, breast tenderness, retention of fluid, nausea, and vomiting).
  Used a 5-point scale ranging from 0 (not at all) to 4 (very much).
  The scores from the 6 estrogen adverse effect items were summed to produce a single score, ranging from 0-24, with higher scores indicating higher adverse effects.
Time Frame: Baseline and Day 28
Population: 27 out of 34 participants in Arm 1 and 22 out of 32 participants in Arm 2 completed both the baseline and Day 28 (4 week) 6 item adverse effect questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 27 | 22
units on a scale
  Baseline | 0.47 (0.48) | 0.46 (0.59)
  Day 28 | 0.70 (0.55) | 0.92 (0.87)

4. Secondary Outcome: Quality of Life (FACT-B Mean Score)
Description: Surveyed using the multidimensional Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire
  The FACT-B (version 4) questionnaire consists of 36 items with five-point scale, ranging from 0-4, where a total score ranges from 0-144 and higher scores indicate better QoL. The total FACT-B score is the sum of scores for five subscales including: physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and specific breast cancer concerns (9 items).
Time Frame: Day 28
Population: 25 out of 34 participants in Arm 1 and 23 out of 32 participants completed the FACT-B questionnaire at Day 28 (4 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 25 | 23
units on a scale | 109.5 (17.9) | 106.9 (21.2)

5. Secondary Outcome: Frequency of Response to Re-treatment With the Same Aromatase Inhibitor That Immediately Preceded Treatment With Estradiol on Protocol.
Description: Best overall response
Time Frame: 12 weeks post-treatment termination
Population: Only offered to patients experiencing clinical benefit on estradiol.
Measure: Number; unit: participants
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 4 | 3
participants
  Partial response | 1 | 1
  Stable disease | 1 | 0
  Progressive disease | 2 | 2

6. Secondary Outcome: Frequency of Response to Re-treatment With Estradiol for Patients Who Have a Secondary Response to an Aromatase Inhibitor After the First Response to Estradiol.
Time Frame: Every 3 months
Population: At the time that the study was powered there was not any information on any patients who were re-treated with estradiol after having a secondary response to a aromatase inhibitor after the first response to estradiol.
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Time Frame: Until patient death
Population: This outcome measure was not analyzed as the overall survival was not reported.
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 0 | 0

8. Post Hoc Outcome: Metabolic Flare on FDG-PET/CT as Compared to Response
Time Frame: Baseline and 24 hours after administration of the first dose of estradiol
Population: The data was combined as the outcome was not based on comparison of the two groups but comparing the overall FDG-PET/CT metabolic flare to the overall responses.
  10 participants were not evaluable because early toxicity prevented response assessment and the PET data was not considered technically adequate or not available in 8 participants.
Measure: Number; unit: participants
Groups:
- Arm 1 (6 mg Estradiol) and Arm 2 (30 mg Estradiol): Arm 1 = 6 mg of estradiol daily (2 mg tid).
  Arm 2 = 30 mg of estradiol. (10 mg tid)
Arm/Group | Arm 1 (6 mg Estradiol) and Arm 2 (30 mg Estradiol)
Number analyzed (Participants) | 46
participants
  Complete response | 0
  Partial response | 3
  Stable disease | 9
  Progressive disease | 3

ADVERSE EVENTS:
Arm/Group | Arm 1 (6 mg Estradiol) | Arm 2 (30 mg Estradiol)
Serious Adverse Events (participants affected / at risk) | 8/34 | 8/32
Other Adverse Events (participants affected / at risk) | 34/34 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (6 mg Estradiol) (N=34) | Arm 2 (30 mg Estradiol) (N=32)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Acute renal failure (Renal and urinary disorders) | 0 | 1
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1
CNS ischemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Eye pain (Eye disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 2 | 0
GI hemorrhage (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutropenia (Investigations) | 0 | 1
Pain (General disorders) | 0 | 1
Perforated viscus (Surgical and medical procedures) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 1 | 0
Vison loss (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Weight loss (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (6 mg Estradiol) (N=34) | Arm 2 (30 mg Estradiol) (N=32)
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Alkaline phosphtase (Investigations) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 14
Ascites (Gastrointestinal disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 18
Breast pain (Reproductive system and breast disorders) | 7 | 13
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Change in libido (Reproductive system and breast disorders) | 3 | 1
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (Cardiac disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dental pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 7
Dizziness (Nervous system disorders) | 6 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspepsia/heartburn (Gastrointestinal disorders) | 9 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Edema (Blood and lymphatic system disorders) | 7 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Fatigue (General disorders) | 22 | 18
Fever (General disorders) | 4 | 2
Groin pain (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 12
Hematuria (Renal and urinary disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 5 | 12
Hirsuitism (Skin and subcutaneous tissue disorders) | 2 | 2
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 5 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolemia (Investigations) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypertriglyceridemia (Investigations) | 6 | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Infection without neutropenia (Infections and infestations) | 5 | 10
Insomnia (Psychiatric disorders) | 10 | 11
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukocytes (Investigations) | 2 | 0
Lymphopenia (Investigations) | 5 | 7
Migraine (Nervous system disorders) | 0 | 2
Mood alteration - anxeity (Psychiatric disorders) | 11 | 5
Mood alteration - depression (Psychiatric disorders) | 5 | 3
Motor neuropathy (Nervous system disorders) | 0 | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 16 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 19 | 16
Neutrophils (Investigations) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Pigmentation change (Skin and subcutaneous tissue disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritis/itching (Skin and subcutaneous tissue disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
SGOT (AST) (Investigations) | 1 | 1
Sensory neuropathy (Nervous system disorders) | 2 | 6
Sinus arrythmia (Cardiac disorders) | 1 | 1
Skin (cellulitis) (Infections and infestations) | 0 | 1
Skin bruising (Skin and subcutaneous tissue disorders) | 1 | 1
Sweating (General disorders) | 0 | 1
Taste alteration (Gastrointestinal disorders) | 1 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Tumor flare - infiltrating tumor in the orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureter pain (Renal and urinary disorders) | 1 | 2
Urinary frequency/urgency (Renal and urinary disorders) | 5 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Vaginal bleeding (Reproductive system and breast disorders) | 7 | 6
Vaginal discharge (Reproductive system and breast disorders) | 7 | 7
Vaginal dryness (Reproductive system and breast disorders) | 2 | 0
Voice change (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 10
Weight gain (Investigations) | 7 | 4
Weight loss (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
The slight imbalance in numbers assigned to the 2 groups was a because of yearly data and safety monitoring, which led to early closure of the 30mg group for toxicity concerns after 32 patients had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes